CLINICAL TRIAL: NCT03866928
Title: Pharmacokinetic Study of Stiripentol and Its Metabolites After Multiple Dose Oral Administration in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STP199
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — stiripentol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stiripentol (Experimental)
  Interventions: Drug: Stiripentol

INTERVENTIONS:
Drug: Stiripentol — 1500 mg of stiripentol b.i.d.

SUMMARY:
This is a monocentric open label study to assess the PK parameters of stiripentol and its metabolites (if any are detected) after multiple oral doses in 14 healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be required to satisfy the following criteria:

1. Healthy male subject, aged between 18 and 45 years inclusive.
2. Considered as healthy after a comprehensive clinical assessment (detailed medical history and complete physical examination).
3. Body mass index (BMI) between 18 and 30 kg/m² inclusive.
4. Normal blood pressure (BP) and heart rate (HR) at the screening visit after 5 min in supine position:

   * 90 mmHg ≤ Systolic Blood Pressure (SBP) ≤ 145 mmHg,
   * 45 mmHg ≤ Diastolic Blood Pressure (DBP) ≤ 90 mmHg,
   * 40 bpm ≤ HR ≤ 90 bpm,
   * Or considered not clinically significant (NCS) by the Investigator.
5. Normal electrocardiogram (ECG) recording on a 10 min resting 12-lead ECG at the screening visit:

   * 120 ≤ interval between P and R waves (PR) < 210 ms,
   * Interval between Q and S waves (QRS) < 120 ms,
   * Fridericia corrected interval between Q and T waves (QTcF) ≤ 450 ms,
   * No sign of any trouble of sinusal automatism,
   * Or considered NCS by the Investigator.
6. Laboratory parameters within the normal range of the laboratory (hematological, blood chemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator.
7. Normal dietary habits.
8. Has given written informed consent.

Exclusion Criteria:

All the subjects included in the study must not meet any of the following non-inclusion criteria.

1. Unsuitable veins for repeated venipuncture.
2. Any relevant history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic, infectious disease or psychiatric disorders,
3. Evidence of any clinically significant acute or chronic disease,
4. Surgery or blood donation (including in the frame of a clinical trial) within 2 months before administration,
5. Presence or relevant history of drug hypersensitivity, asthma or allergic disease diagnosed and treated by a physician,
6. Known hypersensitivity to any of the test materials or related compounds,
7. Inability to abstain from intensive muscular effort,
8. Inability or difficulty swallowing whole capsules
9. No possibility of contact in case of emergency,
10. Any drug intake (except paracetamol) including over the counter (OTC) medications and herbal products that could affect the outcome of the study, within 2 weeks prior to the first drug administration or less than 5 times the t1/2 of that drug, whichever is longer,
11. Who receive carbamazepine, phenytoin or phenobarbital known to affect hepatic metabolism within 1 month prior to the first dose administration,
12. Who receive any drug known to interfere with CYP enzymes within 1 month prior to the first dose administration,
13. History or presence of drug or alcohol abuse (alcohol consumption > 4 glasses per day (1 glass is approximately equivalent to: beer [354 mL], wine [118 mL], or distilled spirits [29.5 mL]) per day)),
14. Excessive consumption of beverages with xanthine bases (> 5 cups or glasses / day),
15. Current use of nicotine containing products, i.e., more than 5 cigarettes or equivalent/day or the inability to stop using nicotine containing products during confinement in the clinical center,
16. Intake of any food or any beverage containing grapefruit or grapefruit juice within one week prior to the first dosing and the inability to stop such intake during the study,
17. Positive Hepatitis B surface antigen (HBsAg) or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests,
18. Positive results of screening for drugs of abuse,
19. Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development,
20. Exclusion period of a previous study,
21. Administrative or legal supervision.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | On Days 1 and 15
  To determine Cmax of stiripentol and its metabolites (if any are detected) in plasma
Area Under the Curve [AUC] | On Days 1 and 15
  To determine AUC of stiripentol and its metabolites (if any are detected) in plasma
Time that a drug is present at the maximum concentration [Tmax] | On Days 1 and 15
  To determine Tmax of stiripentol and its metabolites (if any are detected) in plasma
The minimum concentration [Cmin] | From Day 2 to Day 15
  To determine Cmin of stiripentol and its metabolites (if any are detected) in plasma
Amount of drug excreted in urine [Ae] | From Day 2 to Day 15
  To determine Ae of stiripentol and its metabolites (if any are detected) in urine
Fraction of the dose excreted in urine [fe] | From Day 2 to Day 15
  To determine fe of stiripentol and its metabolites (if any are detected) in urine

SECONDARY OUTCOMES:
Treatment-related adverse events [TRAEs] | From start of participation of the subject until 4 weeks after the last administration of the study drug
  To assess the safety and tolerability of stiripentol and its metabolites (if any are detected) after multiple oral doses of 1500 mg b.i.d in healthy male volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- ATC, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No